CLINICAL TRIAL: NCT06835517
Title: Design of Tools to Transform the Conceptualization of Clinical Error Within and Outside Healthcare Centers, Social-health Centers, Hospitals and Healthcare Management
Brief Title: DECIDE Just Culture: Conceptualization of Clinical Error
Acronym: DECIDE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Collaborators: Hospital Universitario Ramon y Cajal (Other); Hospital Universitario Fundación Alcorcón (Other)
Responsible Party: Principal Investigator, José Joaquín Mira Solves, Dr., Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UGP-24-005; PI24/00243 (Other Grant/Funding Number: ISCIII); PI24/00376 (Other Grant/Funding Number: ISCIII); PI24/00901 (Other Grant/Funding Number: ISCIII)
Record Dates: First submitted 2025-02-06; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Error Disclosure
Keywords: Just Culture; clinical error; honest mistake
MeSH Terms: interventions — Theory of Planned Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Subjects in the control group will participate in a lecture (40 minutes and 15 minutes of discussion) on patient safety, causes of clinical errors and measures to reduce them in healthcare centers.
- Theory of Dissonance (Experimental): This theory describes psychological discomfort when people have thoughts or beliefs that conflict with each other, or when their actions are not aligned with their beliefs or values. In these cases, the intervention seeks this discrepancy by presenting dissonant information, which leads to an adjustment of one's beliefs and attitudes, and thus of one's behaviours.
  Interventions: Behavioral: Theory of Dissonance
- Theory of Reasoned Action (Experimental): This theory provides a conceptual framework for understanding how social norms influence the formation of intentions, and how these intentions predict behaviour. It is especially useful for changing behaviour by modifying the beliefs and norms that underlie attitudes based on the social influence exerted by peers.
  Interventions: Behavioral: Theory of Reasoned Action

INTERVENTIONS:
Behavioral: Theory of Dissonance — The design of this intervention will consist of presenting information that generates dissonance with the subjects' attitudes and beliefs about clinical errors. Dissonance will be intensified by experiential experiences through simulations that provide compelling information that supports the idea of accepting honest errors as learning opportunities within the framework of a Just Culture.
  Arms: Theory of Dissonance
Behavioral: Theory of Reasoned Action — The intervention will consist of the presentation, to the different groups, of testimonies, narratives, statements and analysis of everyday clinical practice situations that promote a change in the so-called "subjective norms" (a person's beliefs about whether significant people in his or her life approve or disapprove of a specific behavior) in relation to the acceptance of honest mistakes (including learning and improving health care from error).
  Arms: Theory of Reasoned Action

SUMMARY:
The main objective of this project is to extend the principles of Just Culture in primary care, hospitals and social-health centers, providing new information on key elements in the social and professional conceptualization of the human factor (fallibility) in safety incidents.

A mixed design combining cross-sectional observational studies based on qualitative (focus groups and consensus conference) and quantitative (survey) methodology with an experimental study or randomized clinical trial with three arms will be used.

The methodology is deployed in four stages or phases of the study:

1. Focus Group technique (qualitative research) with 70 primary care health professionals, 80 hospital health professionals, 70 health professionals from socio-health centers, 72 health managers and 80 social leaders to identify key elements of the subjective norms and social influence processes that define the conceptualization of a clinical error, including impact of gender bias and other stereotypes in relation to blame.
2. Online survey of a stratified random sample of 1,255 managers, middle managers and professionals from primary care, hospitals and social-health centers to analyze the barriers and facilitating factors for the implementation of Just Culture.
3. Randomized experimental study with three arms (84 subjects in each) and control group to determine the effectiveness of two interventions aimed at modifying attitudes, beliefs and behaviors in relation to honest mistakes, based on the Theory of Dissonance and Reasoned Action, both in social leaders and professionals.
4. Application of AGREE II and Consensus Conference technique (33 experts) to elaborate a guide of recommendations in order to implement Just Culture in primary care, with the involvement of all actors (social and professional level) that will be transferred to practice.

DETAILED DESCRIPTION:
Researchers will compare with a control group the effectiveness of two interventions to modify attitudes, beliefs and behaviors in relation to honest mistakes, based on the theory of dissonance and reasoned action, in both social and professional leaders.

The design of intervention A will consist of presenting information that generates dissonance with subjects' attitudes and beliefs about clinical errors. The dissonance will be intensified by experiential experiences through simulations that provide convincing information that supports the idea of accepting honest errors as learning opportunities within the framework of a Just Culture.

The psychoeducational intervention B based will consist of the presentation of testimonials, narratives, statements and analysis of everyday clinical practice situations that promote a change in so-called "subjective norms" (a person's beliefs about whether significant people in their life approve or disapprove of a specific behavior) in relation to the acceptance of honest errors (including learning and improving healthcare from error).

ELIGIBILITY:
Phase 1

* Inclusion criteria: Over 18 years of age, health professionals in primary care, hospitals or social-health centers with more than 5 years of experience. Healthcare managers. People who exercise social leadership in associations, media, blogs, etc. Subjects who voluntarily agree to participate after informed consent and who commit to a dedication of 5 hours.
* Exclusion criteria: Experience in patient safety groups/committees. Ongoing or serious adverse event claims or litigation with institutions.

Phase 2

* Inclusion criteria: Managers of health centers, hospitals or socio-health centers in Andalusia, Aragon, Valencia and Madrid, with a minimum of 7 years of experience, who agree to participate.
* Exclusion criteria:Litigation or claim in the last 15 years.

Phase 3

* Inclusion criteria: Same as in phase 1, who voluntarily agree to participate and commit to a dedication of 90 minutes.
* Exclusion criteria: Same as in phase 1. Who have participated in phase 1.

Phase 4

- Inclusion criteria: Male/female balance, minimum 10 years of experience. Recruitment, among members of SEDISA, SEMERGEN, SEMFyC, FAECAP and other scientific societies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1255 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of attitudes classified as honest mistakes, risky behaviour and reckless behaviour identified in the different video scenarios during the group sessions | 8 months
  The Focus Group technique (face-to-face) will be used to describe the participants' vision of human fallibility. The following will be considered: consistency between contributions (triangulation within and between groups), spontaneity (number of different original contributions); intensity, weighting assigned to each of the ideas (on a scale of 1 to 5 points); and relevance (considering the agreement they arouse by means of the coefficient of variation). Discussions will be held until the information is saturated. In addition, the data collected from the different groups will be triangulated to present joint results.
Number and intensity of the barriers detected that hinder the implementation of Just Culture in the organizations | 11 months
  The Just Culture Assessment Tool (Petschonek et al. J Patient Saf. 2013;9:190-7) and Safety Culture Stack approach (Kirwan et al. Safety and Reliability 2018;38(3):200-217) will be used after cross-cultural adaptation. ANOVA will be used to analyze the relationships between care levels and professional profiles. The t-test statistic will be used to determine differences between men and women. Multiple linear regression will be used taking as dependent variable: scale score and as factors: years of experience, sex, professional profile, autonomous community.
Cost-effectiveness of psychoeducational interventions A and B | 18 months
  Cost-effectiveness will be assessed using a cost-effectiveness analysis, comparing the direct and indirect costs of each intervention with their impact on attitudes, behavioral intention, and cognitive dissonance.
Existence of a guide of recommendations for implementing Just Culture that complies with AGREE II criteria | 8 months
  The Consensus Conference technique will be used to obtain a guide that complies with the AGREE II (Appraisal of Guidelines for Research and Evaluation) principles and that includes recommendations for implementing Just Culture in the different healthcare institutions, adapted to the context.

SECONDARY OUTCOMES:
Behavioral Intention | 18 months
  Measured with an instrument based on the Error-Oriented Motivation Scale and the Safety Attitudes Questionnaire. The best performing items will be selected and their cross-cultural validity and metric properties (according to COSMIN guidelines) will be guaranteed. Assessments at three points in time: before the intervention, at the end of the intervention period and 6 months after.
Cognitive Dissonance | 18 months
  Measured through linguistic indicators of cognitive conflict. Assessments at three points in time: before the intervention, at the end of the intervention period and 6 months later.
Effects of the Intervention | 18 months
  Independently analysed by group using a linear mixed effects model (LMM) for repeated measures. Consideration of data matching and stratification by gender, age, participant profile and intervention arm.

CONTACTS AND LOCATIONS:
Overall Officials: Jose J Mira, Principal Investigator — Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana; Susana Lorenzo Martínez, Principal Investigator — Hospital Universitario Fundación Alcorcón; Jesús M Aranaz Andrés, Principal Investigator — Hospital Universitario Ramón y Cajal
Locations (1):
- Centro de Salud Hospital Plá, Alicante, Spain

REFERENCES:
- [Derived] Mira JJ, Lorenzo S, Aranaz-Andres JM, Macias-Maroto M, Cobos-Vargas A, Moreno Campoy EE, Perez-Perez P, Trillo-Lopez P, Corpas-Nogales E, Gea Velazquez de Castro MT, Arencibia-Jimenez M, Asencio A, Diez Herrero D, Molina-Ribera J, Calderon E, Lozano-Gago P, Libano Beristain A, Navarro Macia C, San Jose Saras D, Gil-Hernandez E, Carrillo I. Understanding and reframing clinical errors through just culture: protocol for the DECIDE mixed-methods study in Spanish healthcare and community contexts. BMJ Open. 2025 Oct 20;15(10):e101421. doi: 10.1136/bmjopen-2025-101421. PMID 41120161